CLINICAL TRIAL: NCT01512979
Title: A 24-week, Randomized, Double-blind, Active-controlled, Parallel Group Trial to Assess the Superiority of Oral Linagliptin and Metformin Compared to Linagliptin Monotherapy in Newly Diagnosed, Treatment-naïve, Uncontrolled Type 2 Diabetes Mellitus Patients
Brief Title: Linagliptin and Metformin Versus Linagliptin in Newly Diagnosed, Untreated Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.83; 2011-004158-24 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Linagliptin

ARMS (2):
- linagliptin (Experimental): patients receive linagliptin tablet once daily
  Interventions: Drug: linagliptin; Drug: metformin placebo
- linagliptin plus metformin (Experimental): patients receive linagliptin tablet once daily and metformin tablets twice daily
  Interventions: Drug: metformin; Drug: linagliptin; Drug: metformin placebo

INTERVENTIONS:
Drug: metformin — 1000 mg to 2000 mg per day
  Arms: linagliptin plus metformin
Drug: linagliptin — 5 mg daily
Drug: metformin placebo — 0 to 2 tablets daily
  Arms: linagliptin plus metformin
Drug: metformin placebo — 4 tablets daily
  Arms: linagliptin

SUMMARY:
The purpose of this trial is to determine whether a initial combination of linagliptin and metformin compared to linagliptin alone for 24 weeks is effective in newly diagnosed, treatment-naïve patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion criteria:

1. Patients must sign and date an Informed Consent consistent with International Conference on Harmonisation / Good Clinical Practice guidelines and local regulations prior to any evaluation and participation in the trial.
2. Male and female patients, 18 years of age or older at Visit 1 (Screen), with newly diagnosed (less than 12 months prior to Screen) Type 2 Diabetes Mellitus.
3. Patients who are treatment-naïve, defined as absence of any oral antidiabetic therapy, injectable glucagon-like peptide-1 agonist/analogue, or insulin, and uncontrolled for the 12 weeks prior to randomisation.
4. Patients must have an glycated (or glycosylated) haemoglobin (HbA1c) between 8.5% [69 millimoles per mole (mmol/mol)] and 12.0% (108 mmol/mol) at Visit 1 (Screen).
5. Patients must have a Body Mass Index (BMI) of 45 kg/m2 or less at Visit 1 (Screen).
6. In the investigators opinion, patients must be reliable, honest, compliant, and agree to cooperate with all planned future trial evaluations as explained in detail during the informed consent process and to be able to perform them.

Exclusion criteria:

Patients with, who are, who have, or who have had:

1. Acute coronary syndrome (non-ST Elevation Myocardial Infarction (STEMI), STEMI, and unstable angina pectoris), stroke or transient ischemic attack within 3 months prior to informed consent.
2. Indication of liver disease determined during Screen and/or Run-In Period, defined by a serum level above 3 times the upper limit of normal (ULN) in any of the following: alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase. Gilbert-Meulengracht syndrome (also known as conjugated hyperbilirubinemia, constitutional hepatic dysfunction, or familial nonhemolytic jaundice) will be permitted.
3. Impaired renal function, defined as calculated creatinine clearance of less than 60 milliliters per minute (< 60 mL/min), by the Cockcroft-Gault Equation, as determined during Screen and/or Run-In Period.
4. Bariatric, gastric bypass, and other gastrointestinal surgeries (including all types of gastric banding and/or LapBand) within the past two years.
5. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
6. Medical history of pancreatitis.
7. Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells (e.g., malaria, babesiosis, haemolytic anaemia).
8. Any contraindication to metformin and/or linagliptin therapies, according to local labels.
9. Treatment with anti-obesity drugs, including over-the-counter drugs such as Alli (orlistat), 3 months prior to informed consent or any other treatment at the time of screening (i.e., surgery, aggressive diet regimen, etc.) leading to unstable body weight.
10. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except Type 2 Diabetes Mellitus.
11. Pre-menopausal women (last menstruation of 1 year or less prior to informed consent) who are nursing or pregnant, are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the trial and do not agree to submit to periodic pregnancy testing during participation in the trial.

    Note: Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems, oral, implantable, intra-vaginal, or injectable contraceptives, Essure micro-inserts placed more than six months prior to Screen Visit, complete sexual abstinence (if acceptable by local authorities), double barrier method (e.g., diaphragm or condom and spermicide), and vasectomised partner.
12. Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance to trial procedures or study medication intake in the opinion of the investigator.
13. Participation in another trial with an investigational drug within 2 months prior to informed consent.
14. Any other clinical condition that would jeopardize patient safety while participating in this clinical trial in the opinion of the Investigator.
15. Inability to commit to regular overnight fasting of at least 10 hours duration and attendance to study site visits between 07:00 and 11:00 ante meridiem (a.m.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (82):
- United States (29):
  - 1218.83.11002 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1218.83.11036 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1218.83.11011 Boehringer Ingelheim Investigational Site, Chino, California
  - 1218.83.11001 Boehringer Ingelheim Investigational Site, Huntington Beach, California
  - 1218.83.11019 Boehringer Ingelheim Investigational Site, Huntington Park, California
  - 1218.83.11015 Boehringer Ingelheim Investigational Site, Lomita, California
  - 1218.83.11023 Boehringer Ingelheim Investigational Site, Norwalk, California
  - 1218.83.11014 Boehringer Ingelheim Investigational Site, Roseville, California
  - 1218.83.11031 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1218.83.11022 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1218.83.11025 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1218.83.11033 Boehringer Ingelheim Investigational Site, Sanford, Florida
  - 1218.83.11029 Boehringer Ingelheim Investigational Site, Oakwood, Georgia
  - 1218.83.11026 Boehringer Ingelheim Investigational Site, Owensboro, Kentucky
  - 1218.83.11008 Boehringer Ingelheim Investigational Site, Elkton, Maryland
  - 1218.83.11027 Boehringer Ingelheim Investigational Site, Freemont, Nebraska
  - 1218.83.11005 Boehringer Ingelheim Investigational Site, Edison, New Jersey
  - 1218.83.11013 Boehringer Ingelheim Investigational Site, Jacksonville, North Carolina
  - 1218.83.11028 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 1218.83.11009 Boehringer Ingelheim Investigational Site, Shelby, North Carolina
  - 1218.83.11003 Boehringer Ingelheim Investigational Site, Franklin, Ohio
  - 1218.83.11024 Boehringer Ingelheim Investigational Site, Gallipolis, Ohio
  - 1218.83.11018 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1218.83.11004 Boehringer Ingelheim Investigational Site, Bristol, Tennessee
  - 1218.83.11017 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1218.83.11032 Boehringer Ingelheim Investigational Site, Grand Prairie, Texas
  - 1218.83.11030 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.83.11034 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.83.11021 Boehringer Ingelheim Investigational Site, Tomball, Texas
- Canada (10):
  - 1218.83.12011 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.83.12007 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1218.83.12001 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1218.83.12002 Boehringer Ingelheim Investigational Site, Paradise, Newfoundland and Labrador
  - 1218.83.12009 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1218.83.12010 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1218.83.12005 Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - 1218.83.12006 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1218.83.12003 Boehringer Ingelheim Investigational Site, Smiths Falls, Ontario
  - 1218.83.12012 Boehringer Ingelheim Investigational Site, Winnipeg, Ontario
- India (3):
  - 1218.83.91003 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.83.91005 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.83.91001 Boehringer Ingelheim Investigational Site, Mumbai
- Israel (3):
  - 1218.83.97004 Boehringer Ingelheim Investigational Site, Haifa
  - 1218.83.97005 Boehringer Ingelheim Investigational Site, Haifa
  - 1218.83.97007 Boehringer Ingelheim Investigational Site, Holon
- Malaysia (3):
  - 1218.83.60001 Boehringer Ingelheim Investigational Site, Kelantan
  - 1218.83.60002 Boehringer Ingelheim Investigational Site, Perak
  - 1218.83.60003 Boehringer Ingelheim Investigational Site, Selangor, Malaysia
- Mexico (5):
  - 1218.83.52004 Boehringer Ingelheim Investigational Site, Cuautla
  - 1218.83.52001 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1218.83.52002 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1218.83.52005 Boehringer Ingelheim Investigational Site, Mérida
  - 1218.83.52003 Boehringer Ingelheim Investigational Site, Tampico
- Philippines (7):
  - 1218.83.63001 Boehringer Ingelheim Investigational Site, Cebu
  - 1218.83.63007 Boehringer Ingelheim Investigational Site, Cebu City
  - 1218.83.63003 Boehringer Ingelheim Investigational Site, Iloilo City
  - 1218.83.63008 Boehringer Ingelheim Investigational Site, Iloilo City
  - 1218.83.63002 Boehringer Ingelheim Investigational Site, Marikina City
  - 1218.83.63006 Boehringer Ingelheim Investigational Site, Marikina City
  - 1218.83.63004 Boehringer Ingelheim Investigational Site, Quezon
- 1218.83.11037 Boehringer Ingelheim Investigational Site, San Juan, Puerto Rico
- Russia (7):
  - 1218.83.07001 Boehringer Ingelheim Investigational Site, Kazan'
  - 1218.83.07002 Boehringer Ingelheim Investigational Site, Petrozavodsk
  - 1218.83.07003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.83.07007 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.83.07004 Boehringer Ingelheim Investigational Site, Samara
  - 1218.83.07006 Boehringer Ingelheim Investigational Site, Smolensk
  - 1218.83.07005 Boehringer Ingelheim Investigational Site, Yaroslavl
- Sri Lanka (4):
  - 1218.83.94004 Boehringer Ingelheim Investigational Site, Dehiwala
  - 1218.83.94002 Boehringer Ingelheim Investigational Site, Galle, Sri Lanka
  - 1218.83.94003 Boehringer Ingelheim Investigational Site, Kandy
  - 1218.83.94001 Boehringer Ingelheim Investigational Site, Ragama
- Thailand (3):
  - 1218.83.66002 Boehringer Ingelheim Investigational Site, Bangkok
  - 1218.83.66003 Boehringer Ingelheim Investigational Site, Bangkok
  - 1218.83.66001 Boehringer Ingelheim Investigational Site, Muang, Khonkaen
- Ukraine (7):
  - 1218.83.38007 Boehringer Ingelheim Investigational Site, Dnipro
  - 1218.83.38001 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 1218.83.38006 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.83.38004 Boehringer Ingelheim Investigational Site, Odesa
  - 1218.83.38008 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1218.83.38003 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 1218.83.38005 Boehringer Ingelheim Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Ross SA, Caballero AE, Del Prato S, Gallwitz B, Lewis-D'Agostino D, Bailes Z, Thiemann S, Patel S, Woerle HJ, von Eynatten M. Linagliptin plus metformin in patients with newly diagnosed type 2 diabetes and marked hyperglycemia. Postgrad Med. 2016 Nov;128(8):747-754. doi: 10.1080/00325481.2016.1238280. Epub 2016 Sep 29. PMID 27684308

RESULTS

PARTICIPANT FLOW:
Groups:
- Linagliptin 5mg + Metformin: Patients treated with linagliptin 5mg and metformin IR (1500mg to 2000mg total daily dose)
- Linagliptin 5mg: Patients treated with linagliptin 5mg
Period: Overall Study
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Started | 159 (Randomised and treated) | 157 (Randomised and treated)
Completed | 140 | 135
Not Completed | 19 | 22
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 1 | 4
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Reason other than stated above | 13 | 9

BASELINE CHARACTERISTICS:
Population: Patients from Treated Set (TS): All patients treated with at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg | Total
Number analyzed (Participants) | 159 | 157 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (10.9) | 48.6 (11.2) | 48.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 80 | 170
  Male | 69 | 77 | 146
Baseline HbA1c [Mean (Standard Deviation); unit: percentage] — Baseline HbA1c was analyzed for the Full Analysis Set which includes all patients randomised, treated with at least 1 dose of study drug, with a baseline HbA1c value and at least 1 on-treatment HbA1c value. The Linagliptin 5mg + Metformin group includes 153 participants, the Linagliptin 5mg group includes 150 participants (303 participants in total).
  percentage | 9.79 (1.19) | 9.88 (1.10) | 9.83 (1.14)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c After 24 Weeks
Description: HbA1c is measured as a percentage. The change from baseline is the Week 24 HbA1c minus the baseline HbA1c. Means are adjusted for treatment and continuous baseline HbA1c
Time Frame: Baseline and 24 weeks
Population: Per Protocol completers cohort (PPCC): All patients randomised, treated with at least 1 dose of study drug, with a baseline HbA1c value without important protocol violations and who completed 24 weeks of treatment, were not treated with rescue medication and have an HbA1c measurement after 24 weeks of treatment.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Number analyzed (Participants) | 132 | 113
percent | -2.81 (0.12) | -2.02 (0.13)
Statistical Analysis 1: Comparison: Linagliptin 5mg + Metformin vs Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — The model includes treatment and continuous baseline HbA1c; Mean Difference (Final Values) = -0.79, 95% CI [-1.13 to -0.46], Standard Error of Mean 0.17

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 24 Weeks of Treatment
Description: The change from baseline is the FPG after 24 weeks minus the baseline FPG. Means are adjusted for treatment, continuous baseline HbA1c and continuous baseline fasting plasma glucose.
Time Frame: Baseline and 24 weeks
Population: Patients from PPCC (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Number analyzed (Participants) | 132 | 113
mg/dL | -47.1 (3.8) | -30.2 (4.2)
Statistical Analysis 1: Comparison: Linagliptin 5mg + Metformin vs Linagliptin 5mg; Test type: Superiority or Other; p = 0.0032, ANCOVA — The model includes treatment, continuous baseline HbA1c and continuous baseline FPG; Mean Difference (Final Values) = -16.9, 95% CI [-28.0 to -5.7], Standard Error of Mean 5.7

3. Secondary Outcome: Change From Baseline in HbA1c by Visit Over Time
Description: HbA1c is measured as a percentage. The change from baseline is the HbA1c over time minus the baseline HbA1c. The model includes treatment, continuous baseline HbA1c in addition to week repeated within patient, week by baseline HbA1c interaction and week by treatment interaction.
Time Frame: Baseline, 6, 12, 18 and 24 weeks
Population: Patients from PPCC (observed cases)
Measure: Mean (Standard Error); unit: percent
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Number analyzed (Participants) | 132 | 113
percent
  Change to week 6 | -1.97 (0.09) | -1.33 (0.10)
  Change to week 12 | -2.69 (0.11) | -1.85 (0.12)
  Change to week 18 | -2.79 (0.11) | -2.01 (0.12)
  Change to week 24 | -2.81 (0.12) | -2.01 (0.13)

4. Secondary Outcome: Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 0.5% After 24 Weeks of Treatment)
Description: The proportion of patients who achieved HbA1c lowering by at least 0.5% after 24 weeks of treatment.The model includes treatment, and continuous baseline HbA1c.
Time Frame: Baseline and 24 weeks
Population: Patients from PPCC. Non-completers considered as failures.
Measure: Number; unit: participants
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Number analyzed (Participants) | 132 | 113
participants | 124 | 92
Statistical Analysis 1: Comparison: Linagliptin 5mg + Metformin vs Linagliptin 5mg; Test type: Superiority or Other; p = 0.0031, Regression, Logistic — The model includes treatment and continuous baseline HbA1c; Odds Ratio (OR) = 3.830, 95% CI [1.573 to 9.328]

5. Secondary Outcome: Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 1.0% After 24 Weeks of Treatment)
Description: The proportion of patients who achieved HbA1c lowering by at least 1.0% after 24 weeks of treatment. The model includes treatment, and continuous baseline HbA1c.
Time Frame: Baseline and 24 weeks
Population: Patients from PPCC. Non-completers considered as failures.
Measure: Number; unit: participants
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Number analyzed (Participants) | 132 | 113
participants | 116 | 82
Statistical Analysis 1: Comparison: Linagliptin 5mg + Metformin vs Linagliptin 5mg; Test type: Superiority or Other; p = 0.0025, Regression, Logistic — The model includes treatment and continuous baseline HbA1c; Odds Ratio (OR) = 2.920, 95% CI [1.458 to 5.849]

6. Secondary Outcome: Occurrence of Treat to Target Efficacy Response (HbA1c <7.0%) After 24 Weeks of Treatment
Description: The proportion of patients who achieved HbA1c below 7.0% after 24 weeks of treatment. The model includes treatment, and continuous baseline HbA1c.
Time Frame: Baseline and 24 weeks
Population: Patients from PPCC. Non-completers considered as failures.
Measure: Number; unit: participants
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Number analyzed (Participants) | 132 | 113
participants | 81 | 45
Statistical Analysis 1: Comparison: Linagliptin 5mg + Metformin vs Linagliptin 5mg; Test type: Superiority or Other; p = 0.0008, Regression, Logistic — The model includes treatment and continuous baseline HbA1c; Odds Ratio (OR) = 2.448, 95% CI [1.453 to 4.123]

7. Secondary Outcome: Change From Baseline in FPG by Visit Over Time
Description: The change from baseline is the FPG over time minus the baseline FPG. Means are adjusted for treatment, continuous baseline HbA1c, continuous baseline FPG in addition to week repeated within patient, week by baseline FPG interaction and week by treatment interaction.
Time Frame: Baseline, 6, 12, 18 and 24 weeks
Population: Patients from PPCC, Observed Cases
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Number analyzed (Participants) | 132 | 113
mg/dL
  Change to week 6 | -52.3 (3.37) | -31.9 (3.67)
  Change to week 12 | -54.1 (3.49) | -30.5 (3.77)
  Change to week 18 | -52.4 (3.20) | -35.4 (3.46)
  Change to week 24 | -47.1 (3.88) | -30.1 (4.16)

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | Linagliptin 5mg + Metformin | Linagliptin 5mg
Serious Adverse Events (participants affected / at risk) | 3/159 | 2/157
Other Adverse Events (participants affected / at risk) | 39/159 | 51/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin 5mg + Metformin (N=159) | Linagliptin 5mg (N=157)
Coronary artery disease (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin 5mg + Metformin (N=159) | Linagliptin 5mg (N=157)
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Urinary tract infection (Infections and infestations) | 10 | 14
Dyslipidaemia (Metabolism and nutrition disorders) | 14 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 20
Headache (Nervous system disorders) | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.